CLINICAL TRIAL: NCT01469754
Title: Coping With Lymphoma to Enhance Adjustment and Reduce Stress in Lymphoma Survivors
Brief Title: Longitudinal Survey Analysis in Lymphoma Survivors
Acronym: CLEAR Stress
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1107011786
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma; Posttraumatic Stress Disorder; Posttraumatic Growth; Coping; Resilience
Keywords: lymphoma; survivors; posttraumatic growth; posttraumatic stress; longitudinal
MeSH Terms: conditions — Lymphoma; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lymphoma Survivors

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a well-documented phenomenon that occurs in cancer survivors. PTSD is known to cause problems with anxiety, depression, and quality of life. Furthermore, there is little treatment available for cancer survivors who suffer from PTSD.

Posttraumatic Growth, however, is a lesser known phenomenon that also occurs in cancer survivors. It is a positive psychological phenomenon that occurs in some people who have suffered a traumatic event--the people who are able to note a "greater appreciation for life", a "stronger relationship with their family/friends," or a "new found level of spirituality" are examples of instances of posttraumatic growth.

Coping with Lymphoma to Enhance Adjustment and Reduce Stress in Survivors (CLEAR Stress) is a study designed to compare the development of PTSD versus the development of Posttraumatic Growth in lymphoma patients at any stage of the cancer experience, regardless of treatment. The hypothesis is that posttraumatic growth, if it is significant, can reduce the impact of PTSD symptoms in the survivor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lymphoma (includes Waldenstrom's Macroglobulinemia)
* Can read/write/understand English without a translator

Exclusion Criteria:

* Currently Hospitalized
* Active Psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lymphoma survivors who have completed initial treatment within the last 3 months
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Growth | Measured at enrollment

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder (PTSD) | Measured at Enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Regina A Jacob, MD, Principal Investigator — WCMC Research Fellow
Locations (1):
- New York Presbyterian/Weill Cornell Center for Lymphoma and Myeloma, New York, New York, United States

REFERENCES:
- See also: WCMC Link to Study Description — http://www.cornellmedicine.org/trials/cancer-and-blood-disorders/lymphoma/coping-with-lymphoma-to-enhance-adjustment-and-reduce-stress-ptsd.html